CLINICAL TRIAL: NCT00082641
Title: 1) Adenovirus p53 Infected DC Vaccine For Breast Cancer, 2) Translation of Biotechnology Into the Clinic
Brief Title: Neoadjuvant/Adjuvant Chemotherapy, Vaccine & Adjuvant Radiation Therapy in p53-Overexpressing Stage III Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0371-02-FB; CDR0000354507 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-01019 (Registry Identifier: CTRP (Clinical Trials Reporting System)); 3P30CA036727-20S1 (NIH)
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive vaccination comprising p53-infected autologous dendritic cells subcutaneously (SC) 1 week after completion of doxorubicin and cyclophosphamide, 1 week after completion of paclitaxel (or after surgery for patients with stage III disease), and at 6 and 12 weeks after completion of radiotherapy (for a total of 4 vaccinations).
  Interventions: Biological: autologous dendritic cell-adenovirus p53 vaccine
- Arm II (Experimental): Patients receive vaccination comprising p53-infected autologous dendritic cells SC at 6, 8, 10, and 12 weeks after completion of radiotherapy.
  Interventions: Biological: autologous dendritic cell-adenovirus p53 vaccine

INTERVENTIONS:
Biological: autologous dendritic cell-adenovirus p53 vaccine — Given subcutaneously on one of two schedules

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Drugs used in chemotherapy, such as doxorubicin, cyclophosphamide, and paclitaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving vaccine therapy before and/or after chemotherapy and radiation therapy may cause a stronger immune response.

PURPOSE: This randomized phase I/II trial is studying the side effects of two regimens of vaccine therapy and to see how well they work in treating women who are receiving neoadjuvant or adjuvant chemotherapy and adjuvant radiation therapy for stage III breast cancer that overexpresses p53.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of two different schedules of vaccination comprising p53-infected autologous dendritic cells in women with p53-overexpressing stage III breast cancer undergoing neoadjuvant or adjuvant chemotherapy and adjuvant radiotherapy.
* Determine the immune response, in terms of humoral and cellular response, in patients treated with these regimens.
* Determine antigen-specific immune responses in patients treated with these regimens.

OUTLINE: This is a randomized, open-label study. Patients are randomized to 1 of 2 treatment arms.

All patients undergo apheresis for the collection of peripheral blood monocytes that are cultured with interleukin-4 and sargramostim (GM-CSF) to produce dendritic cells. The dendritic cells are infected with a recombinant adenoviral vector containing the wild-type p53 gene.

Patients receive doxorubicin IV and cyclophosphamide IV every 2 weeks for 8 weeks (4 courses) followed 2 weeks later by paclitaxel IV every 2 weeks for 8 weeks (4 courses). Patients with stage III disease then undergo surgery. Three weeks after completion of paclitaxel (or after surgery for patients with stage III disease), patients undergo radiotherapy once daily for 6.5 weeks. Patients are then receive vaccine therapy as per the arm to which they were randomized.

* Arm I: Patients receive vaccination comprising p53-infected autologous dendritic cells subcutaneously (SC) 1 week after completion of doxorubicin and cyclophosphamide, 1 week after completion of paclitaxel (or after surgery for patients with stage III disease), and at 6 and 12 weeks after completion of radiotherapy (for a total of 4 vaccinations).
* Arm II: Patients receive vaccination comprising p53-infected autologous dendritic cells SC at 6, 8, 10, and 12 weeks after completion of radiotherapy.

Treatment in both arms continues in the absence of unacceptable toxicity.

Patients are followed at 1 month, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 20-50 patients (10-25 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer meeting the following criteria:

  * Clinically locally advanced disease (stage III) with a primary tumor at least 4 cm by mammogram, ultrasound, or palpation AND/OR palpable axillary nodes larger than 1 cm
  * Planned neoadjuvant chemotherapy
* p53-overexpressing tumor by immunohistochemistry
* Delayed-type hypersensitivity to at least 1 of 3 standard antigens
* Female
* ECOG 0-1
* WBC > 4,000/mm^3
* Platelet count > 100,000/mm^3
* Bilirubin < 2 times upper limit of normal (ULN)
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative
* Creatinine < 2 times ULNHIV negative
* Fertile patients must use effective contraception during and for at least 6 months after study participation

Exclusion Criteria:

* No prior or concurrent autoimmune disorder
* Not pregnant or nursing/negative pregnancy test
* No other concurrent illness that would preclude study participation
* No prior chemotherapy
* No concurrent participation in another therapeutic clinical trial

Ages: 19 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2009-05-01 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Reed, MD, Study Chair — University of Nebraska
Locations (1):
- Eppley Cancer Center, University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject consented to the study voluntarily withdrew consent prior to assignment to an arm, thus only 23 subjects placed in the study arms and are included in the data analysis.
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Customized [Count of Participants; unit: Participants]
  Participant >= 19 years of age | 11 | 12 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Toxicity to the Vaccine
Description: This outcome measure looks at the safety of the vaccine by documenting the number of grade 2, 3, or toxicities experienced by participants related to the vaccine.
Time Frame: 1 week after each vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 11 | 12
Participants | 0 | 0

2. Primary Outcome: Percent of Patients With an Immune Response to p53-infected Autologous Dendritic Cells
Time Frame: Through study completion, an average of 18 months
Measure: Number; unit: percentage of patients
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 11 | 12
percentage of patients | 100 | 53

3. Primary Outcome: Peak Immune Response as Measured by Number of Spots Per Cells
Description: This outcome measure examined the importance of vaccine timing on antigen-specific relative to the primary cytotoxic therapy on the augmentation of antigen specific immune responses by measuring the duration of immune responses of participants
Time Frame: 6 months after last immunization
Population: Due to the low numbers of participants analyze in each arm, 7 participants analyze in the Early vaccine administration 4 participants analyzed in the late vaccine administration the subjects were analyzed together for this outcome.
Measure: Median (Full Range); unit: spots per 300,000 cells
Groups:
- Arm I - Early Vaccine and Arm II - Late Vaccine Administration: Patients receive vaccination comprising p53-infected autologous dendritic cells subcutaneously (SC) 1 week after completion of doxorubicin and cyclophosphamide, 1 week after completion of paclitaxel (or after surgery for patients with stage III disease), and at 6 and 12 weeks after completion of radiotherapy (for a total of 4 vaccinations).
  autologous dendritic cell-adenovirus p53 vaccine: Given subcutaneously on one of two schedules
Arm/Group | Arm I - Early Vaccine and Arm II - Late Vaccine Administration
Number analyzed (Participants) | 11
spots per 300,000 cells | 8.54 [0.09 to 32.5]

ADVERSE EVENTS:
Time Frame: Adverse Events will be collected from the time the subject signs the consent form and ending 4 weeks following the final (typically the fourth) vaccine. For Arm A is approximately 5 months. For Arm B is approximately 6 months.
Arm/Group | Arm I | Arm II
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 5/11 | 1/12
Other Adverse Events (participants affected / at risk) | 6/11 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=11) | Arm II (N=12)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
skin infection (Infections and infestations) | 1 (1) | 0 (0) — cellulitis
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=11) | Arm II (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
platelet count decreased (Investigations) | 0 (0) | 1 (1)
white blood cell decreased (Investigations) | 2 (2) | 2 (3)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) — pneumonia
neutrophil count decreased (Investigations) | 3 (3) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 0 (0) | 1 (1)
skin infection (Infections and infestations) | 0 (0) | 1 (1) — cellulitis
syncope (Nervous system disorders) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes